CLINICAL TRIAL: NCT07360886
Title: Early Detection of Selected Neuropathologies in Motor Vehicle Drivers
Acronym: NeuroDrive
Status: Recruiting | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Sponsor
Other Study IDs: OP JAK ITI VZ 1; CZ.02.01.01/00/23_021/0008829 (Other Grant/Funding Number: Operational Programme Jan Ámos Komenský financed by the European Union (EU) and the State Budget of Czech Republic)
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Parkinson Disease
Keywords: Neurology; Psychology; Traffic psychology; Vienna Test System; Driving abilities
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson disease cohort: PD patients cohort will consist of 100 patients with parkinson disease aged between 18-85 years, with, with a balanced sex distribution to ensure representativeness and reduce gender bias. The target sample size (N = 100) has been chosen to provide adequate statistical power to detect moderate to strong correlations between clinical and paraclinical measures , we also want to distribute patients regularly across all those ages. Participants with premorbid cognitive impairment or those not clinically stable during the study period will be excluded, also participants with a Hoehn and Yahr stage greater than 4 will be excluded.
- Multiple sclerosis cohort: Multiple sclerosis patient cohort will consist of 100 patients with multiple sclerosis. aged between 18-85 years, with, with a balanced sex distribution to ensure representativeness and reduce gender bias. The target sample size (N = 100) has been chosen to provide adequate statistical power to detect moderate to strong correlations between clinical and paraclinical measures , we also want to distribute patients regularly across all those ages. Participants with premorbid cognitive impairment or those not clinically stable during the study period will be excluded also an Expanded Disability Status Scale (EDSS) score above 6.5 will serve as an exclusion criterion.

SUMMARY:
This study aims to develop accessible methods for the early detection of selected neuropathologies in drivers, focusing on multiple sclerosis and Parkinson's disease. The primary objective is to identify clinical tests that correlate with outcomes from the Vienna Test System (VTS), thereby enabling early diagnosis without the need for complex neurological or neuropsychological assessments. Findings could improve the effectiveness of routine driver medical check-ups and inform future modifications to Czech traffic law to enhance road safety.

DETAILED DESCRIPTION:
The study will be conducted in two phases. First, a cohort of healthy participants will undergo assessment using the Vienna Test System (VTS). Subsequently, a clinical cohort comprising individuals diagnosed with multiple sclerosis (MS) or Parkinson's disease (PD) will be recruited. Each clinical participant will complete a basic neurological examination, including the Montreal Cognitive Assessment (MoCA), 25-Foot Walk Test (25-FWT), Symbol Digit Modalities Test (SDMT), and Nine-Hole Peg Test (9-HPT). They will then undergo VTS testing.

Patients with PD will be classified according to the Hoehn and Yahr scale, while those with MS will be staged using the Expanded Disability Status Scale (EDSS). The aim is to determine which easily accessible clinical tests show the strongest correlation with VTS outcomes, thereby identifying reliable markers that can be incorporated into standard medical evaluations of drivers.

In the second phase, paraclinical findings obtained outside the scope of this study will be used to strengthen the evidence base. Ultimately, the project seeks to propose a risk equation in the form of a practical calculator that physicians can use when evaluating a patient's fitness to drive. An additional anticipated outcome is the development of targeted cognitive and motor training interventions to help drivers with neuropathologies maintain or improve safe driving abilities.

ELIGIBILITY:
Inclusion Criteria:

* Person after signing informed consent.
* After meeting the valid diagnostic criteria for the given neurological diagnosis.
* Possession of a valid driver's license and proof of active driving.
* Age limit 18 - 85 years.

Exclusion Criteria:

* Proven diagnosis of dementia based on a current psychological examination (MMSE 24 points or less).
* Diagnosis of a disease or condition that, according to Czech Law. No. 277/2004 Coll., on medical fitness to drive motor vehicles, as amended (especially Law No. 204/2025 Coll.), prevents or significantly limits the ability to drive a motor vehicle safely (e.g. dementia, epilepsy, severe disorders of consciousness).
* Age less than 18 years.
* Age more than 85 years.
* In the second cohort (patients with Multiple Sclerosis), proven and treated relapse in the last 6 weeks before inclusion in the study.
* In the MS cohort, current EDSS > 6.5 points.
* For the PD cohort, the current Hoehn and Yahr scale score is greater than or equal to 4.
* For both cohorts, evidence of parainfectious deterioration as demonstrated by laboratory testing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the dispensary care of the neurological department of the University hospital Olomouc with the full access to the paraclinical data and demographic features.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Vienna Test Systems (VTS) - Determination Test (DT) | 10 minutes
  Vienna Test System (VTS) - Determination Test (DT). A computerized test of attention, stress tolerance, and psychomotor reactivity under complex conditions. Participants are presented with rapidly changing visual and auditory stimuli (e.g., colored lights, acoustic signals) and must respond as quickly as possible using multiple response keys or pedals.
  Scoring: outcomes include mean and median reaction time (ms), number of correct responses, omission errors (missed stimuli), commission errors (incorrect responses), and measures of performance stability across the task. Faster, more accurate, and stable performance indicates better attentional control and stress tolerance.
  Administration: conducted in a quiet environment with standardized VTS hardware and software. Trained staff provide uniform instructions and monitor performance.
Vienna Test Systems (VTS) - Reaction Test (RT) | 10 minutes
  Vienna Test System (VTS) - Reaction Test (RT). A computerized assessment of simple and choice reaction time measuring perceptual speed and motor response. Participants are presented with visual and/or auditory stimuli and instructed to respond as quickly as possible by pressing a button (simple RT) or selecting the correct response among multiple options (choice RT).
  Scoring: main outcomes include mean reaction time (ms), number of correct responses, and error rates. Faster and more accurate responses indicate better psychomotor speed and attention. Separate scores are calculated for simple and choice conditions.
  Administration: conducted individually in a quiet, distraction-free environment using standardized VTS hardware and software. Trained staff provide standardized instructions and supervise.
Vienna Test Systems (VTS) - Response inhibition (INHIB) | 15 minutes
  Vienna Test System (VTS) - Response Inhibition (INHIB). A computerized go/no-go paradigm measuring impulse control and inhibitory executive function. Participants are presented with a continuous sequence of visual stimuli on screen. They are instructed to respond via button press to "go" stimuli and withhold responses to "no-go" stimuli.
  Scoring: main outcomes include reaction time to go-stimuli, number of correct responses (hits), commission errors (responses to no-go stimuli), and omission errors (missed go-stimuli). Higher accuracy with fewer commission errors reflects better inhibitory control.
  Administration: conducted individually in a distraction-free environment using standardized VTS software and response panel. Trained staff provide instructions and supervise performance.
Vienna Test Systems (VTS) - Vigilance/Sustained attention (WAFV) - Short version | 20 minutes
  Vienna Test System (VTS) - Vigilance/Sustained Attention (WAFV). A computerized test measuring sustained attention and vigilance. Participants monitor a continuous sequence of simple visual stimuli (e.g., small changes in geometric figures) presented at regular intervals. They are instructed to respond via button press whenever a predefined critical stimulus appears.
  Scoring: main outcomes include number of correct detections (hits), omissions (missed targets), false alarms (incorrect responses), and reaction times. Higher hits and faster, stable reaction times indicate better vigilance; higher omissions or false alarms indicate poorer sustained attention.
  Administration: conducted individually in a distraction-free environment using the standardized VTS software and response panel. Trained staff provide instructions and supervise.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 15 minutes
  Montreal Cognitive Assessment (MoCA). A clinician-administered screening tool for mild cognitive impairment covering multiple domains: attention, concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The test consists of 30 items with a maximum total score of 30; higher scores = better cognition. A score of 26 or above is considered normal. If the participant has ≤12 years of formal education, +1 point is added.
  Administration: conducted face-to-face in a quiet environment by trained staff using validated language versions; completion requires ~10-15 minutes.
  Outcomes: total score and change from baseline.
25-Foot Walk Test (25-FWT) | 2 minutes
  25-Foot Walk Test (25-FWT). A quantitative measure of ambulatory function and walking speed. Participants are instructed to walk 25 feet (7.62 m) as quickly and safely as possible. Two trials are performed, typically with a short rest interval, and the average time (in seconds) is recorded using a stopwatch. Lower times = better mobility. Use of customary assistive devices (e.g., cane, walker) is permitted and documented.
  Administration: conducted in a straight, unobstructed corridor with clearly marked start and finish lines. Trained staff provide standardized instructions and supervise for safety. Completion typically requires ~5 minutes.
  Outcomes: average time to walk 25 feet (7.62 meters), ability to complete the test, and change from baseline.
Symbol Digit Modalities Test (SDMT) | 2 minutes
  Symbol Digit Modalities Test (SDMT). A brief neurocognitive test of attention, processing speed, and visual scanning. Participants are shown a key pairing nine symbols with digits 1-9. Using this key, they write or orally state the digit corresponding to each symbol in a randomized sequence presented on the test form.
  Scoring: the number of correct substitutions completed in 90 seconds is counted. Higher scores = better cognitive performance. Errors are recorded but not included in the raw score. Written and oral versions are available; the same mode is used across visits for consistency.
  Administration: conducted in a quiet environment with standardized instructions, requiring ~5 minutes. Staff monitor to ensure task adherence.
  Outcomes: total correct substitutions and standard deviation change from the normal value.
Nine-Hole Peg Test (9-HPT) | 5 minutes
  Nine-Hole Peg Test (9-HPT). A standardized test of finger dexterity and fine motor function. Participants are instructed to place nine pegs into nine holes on a board, one at a time, as quickly as possible, and then remove them. Each hand is tested separately, typically with the dominant hand first, followed by the non-dominant hand.
  Scoring: performance time (in seconds) for each hand is recorded with a stopwatch. Lower times = better dexterity. Two consecutive trials per hand are averaged. If a peg is dropped, the participant retrieves it and continues.
  Administration: administered in a quiet environment by trained staff using standardized instructions. Completion time is usually 3-5 minutes for both hands.
  Outcomes: mean completion time for each hand and change from baseline.
Benton Visual Retention Test (BVRT) | 20 minutes
  A neuropsychological assessment of visual memory, perception, and visuoconstructive ability. Participants are shown a series of 10 geometric designs, each displayed for 10 seconds, and then asked to reproduce the design from memory using paper and pencil (Administration A). Alternate forms may be used to minimize practice effects.
  Scoring: each reproduction is scored for number correct (maximum = 10) and for errors (e.g., omissions, distortions, rotations, perseverations, misplacements). Higher correct scores indicate better performance, while higher error counts indicate impairment.
  Administration: conducted individually in a quiet setting by trained staff; typical completion ~15 minutes.
  Outcomes: total correct responses, total errors, and change from baseline.
The Big Five Inventory-2 Short Form (BFI-2-S) | 15 minutes
  Big Five Inventory-2 Short Form (BFI-2-S). A 30-item self-report assessing five personality domains: Extraversion, Agreeableness, Conscientiousness, Negative Emotionality, and Open-Mindedness. Items are rated on a 5-point Likert scale (1 = disagree strongly to 5 = agree strongly). For each domain, compute the mean of its 6 items after applying the manual's reverse-keying rules; higher scores = more of that trait. No total score is used.
  Administration: validated language version via paper or secure ePRO; typical completion ~5-7 min. Staff provide standardized instructions and check completeness.
  Outcomes: domain scores (1-5) and change from baseline. Timing: baseline and follow-ups within ±3 days of the visit window.
Epworth Sleepiness Scale (ESS) | 5 minutes
  An 8-item self-report of daytime sleepiness. Participants rate their chance of dozing in common situations from 0 (would never doze) to 3 (high chance). Total score = sum of items (range 0-24; higher = worse sleepiness). Severity bands: 0-5 normal, 6-10 higher-than-normal, 11-12 mild, 13-15 moderate, 16-24 severe.
  Administration: validated language version via paper or secure ePRO; typical completion ~2-3 min. Staff provide standardized instructions and check completeness before scoring.
  Outcomes: total score; change from baseline; response = ≥3-point reduction from baseline; remission = score ≤10.
Beck's Depression Inventory (BDI-II) | 8 minutes
  A 21-item self-report questionnaire assessing depressive symptoms over the past 2 weeks, including today. Each item is rated 0-3; total score ranges 0-63, with higher scores indicating more severe depression. Severity categories: 0-13 minimal, 14-19 mild, 20-28 moderate, 29-63 severe. The BDI-II is administered in validated language versions on paper or secure ePRO, requiring ~5-10 minutes. Staff provide standardized instructions and check completeness. Outcomes include total score, change from baseline, response (≥50% reduction from baseline), and remission (score ≤13).
Driving experience self-evaluation questionnaire | 10 minutes
  This self-report questionnaire captures recent driving exposure and perceived difficulties over the past month. Items use 7-point Likert scales anchored "Never (1)" to "Every drive (7)". Content includes deliberate avoidance of challenging conditions (night driving, heavy traffic, bad weather, highways, unfamiliar routes), fatigue while driving, uncertainty in traffic situations (e.g., speed limits, lane selection, right of way), perceived complexity/overload, inattention, vehicle-control errors (e.g., wrong gear, pedal mix-ups), oversight errors (e.g., missed lights/signs, failure to check mirrors), warnings from other road users, risk-taking, traffic-rule violations, and emotional arousal during driving. A brief exposure module records typical driving frequency, lifetime kilometers, and the frequency of driving in specific conditions. Higher scores indicate more frequent difficulties; the primary metric is the mean item score (1-7).

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Olomouc, Olomouc, Olomoucký kraj, Czechia

IPD SHARING:
Plan to Share IPD: No